CLINICAL TRIAL: NCT02663752
Title: A Phase II Pilot Study to Assess the Presence of Molecular Factors Predictive for Hematologic Response in Myelodysplastic Syndrome Patients Receiving Deferasirox Therapy in Hematological Centers in Belgium Using Gene Expressing Profiling From Baseline Bone Marrow.
Brief Title: A Phase II Pilot Study to Assess the Presence of Molecular Factors Predictive for Hematologic Response in Myelodysplastic Syndrome Patients Receiving Deferasirox Therapy.
Acronym: EXPHAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CICL670ABE04
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Myelodysplastic Syndrome
Keywords: deferasirox; MDS; RNA expression; predictive biomarker
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox (Other): All patients are already on commercial deferasirox before entering the study.
  Interventions: Procedure: Bone marrow aspirate; Drug: Deferasirox

INTERVENTIONS:
Procedure: Bone marrow aspirate — Patients experiencing a hematological response and patients not experiencing a hematological response while on deferasirox treatment received a new bone marrow aspirate in order to investigate the presence of differential gene expression between those two groups
Drug: Deferasirox — Patients are already on commercial deferasirox before entering the study.

SUMMARY:
Several previous studies (clinical and non-clinical) hypothesize that treatment with deferasirox causes a hematological improvement in transfused patients with low and intermediate-1 risk myelodysplastic syndrome. The purpose of this study was to assess the presence of genetic biomarkers predictive for hematologic response by the use of gene expression profiling of bone marrow aspirates obtained from MDS patients with or without hematological response.

DETAILED DESCRIPTION:
This trial was terminated due to low enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any other study procedure,
* Males or females ≥ 18 years of age,
* MDS according to WHO criteria lasting ≥ 14 weeks at the time of screening, IPSS score <1.5 (low and intermediate-1 risk patients) at the time of screening using the IPSS score of 1997
* Treatment with deferasirox:
* Only for the responder group: Treatment with deferasirox for prevention or treatment of IOL for at least 14 weeks before screening.
* Only for the non-responder group: Treatment with deferasirox for at least 9 months for prevention or treatment of IOL before screening to exclude patients with a late hematological response.
* Only for responder-group: Patient with hematological response defined according to the IWG criteria of 2006 which must last at least 8 weeks, confirmed by the scientific advisory committee. In case a hematological response is identified retrospectively, the confirmation will be based on the last available blood result showing hematological response according to the IWG criteria of 2006. In this case, an archived bone marrow sample at the moment of response has to be available in order to be eligible. This archived bone marrow had to be taken at the moment when hematological response was present for at least 8 weeks and was still ongoing at the moment of sampling, according to the IWG criteria of 2006 in order to be eligible. When a bone marrow sample was taken after the hematological response had already disappeared, the sample is not eligible for further analysis.
* Only for non-responder group: confirmation by the scientific advisory committee that patient is eligible based on matched-pairing and confirmation of no hematological response. Minimal requirements for matched pairing include age, sex, IPSS score, hemoglobin level, transfusion need at baseline, treatment duration with deferasirox and time since MDS diagnosis. Pairing can be extended according to level of leukopenia, thrombocytopenia, serum ferritin level at baseline, comorbidities and transfusion history. More details about pairing are described in the protocol. In case a non-responder is identified retrospectively and an archival bone marrow is available at that documented time of non-response, this can be used for further analysis. In that case, an interval of 4 weeks between blood sampling for documentation of non-response and bone marrow sampling is allowed.
* Bone marrow aspirate/RNA taken at the time of MDS diagnosis (at baseline) retrievable from patient's hospital. This should be checked by the treating hematologist/oncologist before referring the patient for potential inclusion to the study. This aspirate/RNA has to be preserved under the right circumstances in order to ensure the quality of the RNA. The sample most be frozen viably, meaning controlled rate freezing and addition of a protector dimethyl sulfoxide DMSO and preserved in -80°C. Preservation of cells that are lysed in a lysis buffer upon arrival in the lab, and stored at -20°C until RNA-extraction are also useful for this study.

Exclusion Criteria:

* Known concomitant presence of anemia due to iron, B12 or folate deficiencies, auto-immune or hereditary hemolysis, gastro-intestinal bleeding or medication induced anemia at the time of screening,
* Known infection with viral hepatitis B (HBV) or viral hepatitis C (HCV) defined as the presence in blood of HBV antigens in absence of HB antibodies, or presence of HCV antibodies at the time of screening,
* Known history of positivity to human immunodeficiency virus (HIV) measured by enzyme-linked immunosorbent assay (ELISA) or western blot at the time of screening,
* Patient participating in another clinical trial or receiving any investigational drug at the time of screening within 1 month prior to study inclusion
* History of other malignancy within the last five years, with the exception of basal skin carcinoma or cervical carcinoma in situ or completely resected colonic polyps carcinoma in situ
* Concomitant treatment with other drugs known or suspected to elicit hematological response. (azacitidine, hematopoietic growth factors, granulocyte colony stimulating factors, valproate, lenalidomide, thalidomide, ATG, cyclosporine, arsenic trioxide).When patients are still receiving red blood cell transfusions, patients are still eligible for study inclusion as long as they meet the IWG criteria of 2006
* Female patients who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study has been discontinued because of low patient recruitment.
Period: Overall Study
Arm/Group | Deferasirox
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Due to low recruitment (1 patient after 12 months of recruitment) the study has been cancelled. Because there was only 1 patient who enrolled, it's best that the baseline characteristics of this patient be kept confidential, respecting the privacy of this patient.
Arm/Group | Deferasirox
Number analyzed (Participants) | 0
Age, Customized [unit: years]
Sex/Gender, Customized [unit: number]

OUTCOME MEASURES:

1. Primary Outcome: Fold Increase/Decrease in Gene Transcription From Baseline Bone Marrow Aspirate of Responders Versus Non-responders'
Description: Using next-generation sequencing, gene expression profiling in responder and non-responder patients were to be performed on existing bone marrow aspirate samples. Gene transcription were then to be compared between the two groups and the fold increase/decrease in differentially expressed genes were to be calculated.
Time Frame: 18 months
Population: There was no treatment administration specific to this study. The trial was terminated due to low enrollment. Because of the limited number of data collected an efficacy analysis was not possible.
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Response
Description: The time to response is defined as the time (in months) between the date of deferasirox initiation and the date of the first documented hematological response only in the responder group.
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Serum Ferritin Levels
Description: From baseline to time of response (responder group) or time to last follow up (non-responders)
Time Frame: Baseline, 18 months
Population: as for outcome 1
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

4. Secondary Outcome: Deferasirox Dose Used
Description: Deferasirox dose is defined as the average daily dose (mg/kg/d) given to the patient from treatment initiation to the emergence of hematological response in the responder group or the time of enrollment in the study in the non-responder group.
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Serum Transferrin Levels
Description: From baseline to time of response (responder group) or time to last follow up (non-responders)
Time Frame: Baseline, 18 months
Population: as for outcome 1
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Transferrin Saturation Levels
Description: From baseline to time of response (responder group) or time to last follow up (non-responders)
Time Frame: Baseline, 18 months
Population: as for outcome 1
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Description: There was no treatment administration specific to this study. The trial was terminated due to low enrollment. The patient did not experience any Adverse Events during the trial.
Arm/Group | Deferasirox
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The trial was terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data form all sites) in the clinical trial.